CLINICAL TRIAL: NCT03270631
Title: Movement Control Exercises and Fascial Manipulation in Chronic Low Back Pain in Conjunction With Multidisciplinary Rehabilitation - a RCT
Brief Title: Movement Control Exercises and Fascial Manipulation in Chronic Low Back Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: Loisto Terveys, Oulu (Unknown); Fysios Kastelli, Oulu (Unknown); Faskia-Markus, Oulu (Unknown)
Responsible Party: Principal Investigator, Jani Takatalo, Resident of PRM, PhD, MD, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM&KCStudy
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain; Low Back Pain, Recurrent
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Five groups: 1) control, 2) fascial manipulation (FM) + movement control exercise (MCE), 3) FM + sham-MCE, 4) MCE + sham-FM and 5) sham-FM and sham-MCE
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant are not aware which treatment and exercises they will have, physical therapist who perform treatments and exercise prescription were blinded for measurements and each others work. Outcome assessor was blinded for baseline study results and treatment groups. Investigator was blinded for all the work done by others.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control (No Intervention): Multidisciplinary rehabilitation, no interventions
- FM and MCE (Experimental): Subjects will have 4-5 times of fascial manipulation (FM) treatment and 4-6 times movement control exercises (MCE) at home to be done based on movement control testing (MCT). Both are given in 3 month period.
  Interventions: Other: FM and MCE
- FM and sham-MCE (Other): FM 4-5 times in 3 months and 4 general exercise prescription.
  Interventions: Other: FM and sham-MCE
- MCE and sham-FM (Other): Sham-FM 4 times in 3 months including trigger point treatment in before decided points and 4-6 times MCE prescription and home exercises.
  Interventions: Other: MCE and sham-FM
- Sham-MCE and sham-FM (Sham Comparator): 4 general practice guiding and Sham-FM 4 times in 3 months including trigger point treatment in before decided points.
  Interventions: Other: Sham-MCE and sham-FM

INTERVENTIONS:
Other: FM and MCE — Treatments (FM and MCE) are given individually and as in a normal clinical physical therapy setting.
  Arms: FM and MCE
Other: FM and sham-MCE — Treatments (FM) are given individually and as in a normal clinical physical therapy setting. Sham-MCE is general exercises.
  Arms: FM and sham-MCE
Other: MCE and sham-FM — Treatments (FM and MCE) are given individually and as in a normal clinical physical therapy setting. Sham-FM is similar to trigger point treatment with treated points randomized.
  Arms: MCE and sham-FM
Other: Sham-MCE and sham-FM — Sham-FM is similar to trigger point treatment with treated points randomized. Sham-MCE is general exercises.
  Arms: Sham-MCE and sham-FM

SUMMARY:
Subjects are recruited from the attendees of the multidisciplinary low back pain rehabilitation group before it takes place in University Hospital of Oulu at Physical and Rehabilitation Medicine (PRM) unit. Subjects were invited to participate by letter 2 weeks before the beginning of the rehabilitation. Subjects to rehabilitation are picked by doctor at PRM unit. The volunteered subjects are invited to the briefing of the study and those who are willing to participate, they filled in several questionnaires about pain, participation, disability and mood. After that the subjects are measured at baseline measurement. Subjects are randomized into the five groups. After the 3 months treatment and training the follow-up measurements are performed. Same questionnaires are filled in at that point as well. At 6 and 12 months the follow-up questionnaires (same as before) are sent to subjects.

DETAILED DESCRIPTION:
Subjects are recruited from the attendees of the multidisciplinary low back pain rehabilitation group before it takes place in University Hospital of Oulu at Physical and Rehabilitation Medicine (PRM) unit. Subjects were invited to participate by letter 2 weeks before the beginning of the rehabilitation. Subjects to rehabilitation are picked by doctor at PRM unit. The volunteered subjects are invited to the briefing of the study and those who are willing to participate, they filled in several questionnaires about pain, participation, disability and mood. After that the subjects are measured at baseline measurement. Subjects are randomized into the five groups: 1) control group, 2) fascial manipulation (FM) and movement control exercises (MCE), 3) sham-FM and MCE, 4) FM and sham-MCE and 5) sham-FM and sham-MCE. Physical therapists who perform treatments (FM), prescribing MCE and performing the measurements are blinded to each other. Physical therapist who is performing measurements is also blinded for the baseline measurements. There and 4 treatments of sham-FM, 4-5 treatments of FM, 4 treatments of sham-MCE and 4-6 treatments of MCE. Control group will receive only university hospital rehabilitation and will participate into the baseline and follow-up measurements. After the 3 months treatment and training the follow-up measurements are performed. Same questionnaires are filled in as at baseline. At 6 and 12 months the follow-up questionnaires (same as before) are sent to subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-operatively treated low back pain or pain after the low back operation. Participation in multidisciplinary rehabilitation at University Hospital of Oulu.

Exclusion Criteria:

* Specific low back pain cause and earlier fascial manipulation treatment given.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Specific Functional Scale (PSFS) | Baseline, 3, 6 and 12 months
  Three different meaningful tasks will be rated from 0 to 10 as how hard is the task.

SECONDARY OUTCOMES:
Change in Oswestry | Baseline, 3, 6 and 12 months
  Disability index
Change in PROMIS | Baseline, 3, 6 and 12 months
  Quality of life
Change in Tampa Scale of Kinesiophobia | Baseline, 3, 6 and 12 months
  Fear of movement
Change in Visual analogue Scale | Baseline, 3, 6 and 12 months
  Pain scale
Change in Linton Örebro | Baseline, 3, 6 and 12 months
  Psychosocial risk factor
Change in Start back | Baseline, 3, 6 and 12 months
  Screening tool of the psychosocial risk factors
Change in Movement control tests | Change from baseline at 3 month
  Clinical tests for LBP
Change in Spinal mouse | Change from baseline at 3 month
  Mobility of the spine
Change in Balance measured with computer | Change from baseline at 3 month
  Power plate
Change in Mobility of the hips | Change from baseline at 3 month
  Hip ROM
Change in Two-point discrimination | Change from baseline at 3 month
  How far apart subject is able to feel two distinctive point of touch
Change in Lef-right discrimination | Change from baseline at 3 month
  How subject is able to understand right and left of the back
Change in Ultrasound of the fascia | Change from baseline at 3 month
  Several fascial structures are measured

CONTACTS AND LOCATIONS:
Overall Officials: Jani Takatalo, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- University Hospital of Oulu, Oulu, Finland